CLINICAL TRIAL: NCT03214900
Title: Evaluation of Vascular Regeneration After a Drug Eluting Stent Implantation and the Development of Neointimal Hyperplasia and Stent Restenosis (REVER Trial).
Brief Title: Evaluation of Vascular Regeneration After a Drug Eluting Stent Implantation
Acronym: REVER
Status: Completed | Type: Observational
Sponsor: Hospital San Carlos, Madrid (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Pilar Jimenez Quevedo, MD, PhD, Principal Investigator, Hospital San Carlos, Madrid
Other Study IDs: PI11/00299
Record Dates: First submitted 2017-06-25; First posted 2017-07-12 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Stable Angina
MeSH Terms: conditions — Angina, Stable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective cohort, one center. twenty patients who will undergo percutaneous stent implantation with everolimus eluting stent will be include. The primary endpoint was the correlation between the change (baseline vs. 1 week) in the number of circulating endothelial progenitor cells and in cell functionality following an everolimus eluting stent implantation with the grade of neointimal hyperplasia measured by optical coherence tomography

DETAILED DESCRIPTION:
For the purpose of the study, flow cytometry analyses will be performed before intervention, at 1 week, 1 month and 9 months. In addition, cell functionality analyses will be performed by quantification of colony forming units, aldehidrodehidrogenase activity, cell proliferation by WST-1 and senescence by !-galactosidase enzyme. At 9 months the degree of neointimal proliferation will be measured by optical coherence tomography . A clinical follow-up will be performed at 1 year. Secondary endpoints include: 1. to correlate the change in the number and cell functionality of circulation progenitor cells following everolimus eluting stent and the injury score analyses measured by optical coherence tomography, and the percentage of non covered struts by optical coherence tomography at 9 months.

2.-. To evaluate the role of other subtypes of cells CD 133+/Kinase Insert Domain Receptor (KDR+), CD 14+, mesenchymal stem cells, endothelial cell markers (VE cadherina, P1H12), integrin expression of Macrophage-1 antigen (MAC-1) and the development of neointimal hyperplasia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present stable angina, silent ischemia or unstable angina whenever there is no elevation of markers of myocardial damage above the limit of normality
* Presence of at least one severe coronary stenosis (> 70% by visual analysis), susceptible of percutaneous treatment with stent implantation and an optical coherence Tomography study
* All patients should be taking statins at least 2 months prior to their inclusion in the study.

Exclusion Criteria:

* Age under 18 years and pregnant or fertile age,
* Patients with ST-elevation myocardial infarction or non-ST-elevation acute coronary syndrome with markers of recent myocardial damage (<3 months),
* Patients in whom a drug-eluting stent and a bare stent have been implanted in the same procedure.
* Percutaneous treatment of restenotic lesions or total chronic occlusions.
* The use of stent pre-implantation ablation techniques (rotablator, directional atherectomy).
* Chronic renal insufficiency with serum creatinine greater than or equal to 2.5.
* Coronary revascularization in previous 3 months.
* Severe ventricular dysfunction (<25%).
* Major trauma or surgery in the previous 3 months.
* Previous organ transplantation, active neoplastic process or inflammatory disease, treatment with immunosuppressors.
* Contraindication or allergy to thienopyridines.
* Life expectancy less than one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stable angina
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-07-01 (Actual); Primary Completion 2014-07-01 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
The correlation between the change (baseline vs 1 week) of circulating with neointimal hyperplasia endothelial progenitor cells and in cell functionality following an Everolimus eluting stent implantation with the grade of neointimal hyperplasia | 9 months
  Correlation between the change (baseline vs 1 week) in the number of circulating endothelial progenitor cells and in cell functionality following an everolimus eluting stent implantation with the grade of neointimal hyperplasia measured by optical coherence Tomography

SECONDARY OUTCOMES:
to correlate number of cell and functionality of progenitor cells and injury score following everolimus eluting stent | baseline
  to correlate the number and cell functionality of progenitor cells following everolimus eluting stent and the injury score analyses measured by optical coherence tomography
to evaluate other subtypes of cells with neointimal hyperplasia | 9 months
  To evaluate the role of other subtypes of cells CD 133+/KDR+, following an everolimus eluting stent implantation with the grade of neointimal hyperplasia measured by optical coherence Tomography
to evaluate other subtypes of cells with neointimal hyperplasia | 9 months
  the role of other subtypes of cells CD 14+ following an everolimus eluting stent implantation with the grade of neointimal hyperplasia measured by optical coherence Tomography
to evaluate endothelial cell markers with neointimal hyperplasia | 9 months
  the role of endothelial cell markers (VE cadherin, P1H12) following an everolimus eluting stent implantation with the grade of neointimal hyperplasia measured by optical coherence Tomography
to evaluate integrin expression of MAC-1 (Macrophage-1 antigen) with neointimal hyperplasia | 9 months
  the role of integrin expression of MAC-1(Macrophage-1 antigen) following an everolimus eluting stent implantation with the grade of neointimal hyperplasia measured by optical coherence Tomography

IPD SHARING:
Plan to Share IPD: No